CLINICAL TRIAL: NCT02044094
Title: A Multiple-Dose Study of Blockade of Subjective Opioid Effects, Plasma Levels, and Safety of Subcutaneous Injections of Depot Buprenorphine (RBP-6000) in Subjects With Opioid Use Disorder
Brief Title: Multiple Dose Study of Blockade of Opioid Effects by Injections of Buprenorphine in Participants With Opioid Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-13-0002
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Opioid Use Disorder
Keywords: Opioid dependent; Buprenorphine; Suboxone Film; Opioid blockade; Hydromorphone challenge
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination; Hydromorphone; Saline Solution

STUDY DESIGN:
Intervention Model Description: All subjects were dispensed the same 300 mg dose of the investigational drug, RBP-6000. They were all also exposed to 0 mg, 6 mg, and 18 mg of hydromorphone for challenges sequentially in a randomized manner.
Masking Description: The investigational drug, RBP-6000, was administered unblinded. The hydromorphone challenges used to measure the effectiveness of RBP-6000 were known and randomized in blinded fashion only to determine the order in which they were administered, with participant and clinical staff blinded to the order of dosing.
Oversight: Data Monitoring Committee: No

ARMS (1):
- depot buprenorphine (Experimental): Participants were treated with RBP-6000 300-mg in a single subcutaneous injection on Days 1 and 29 following a prior 14 day stabilization period (day -14 to day -1) of buprenorphine and naloxone (SUBOXONE) . Challenges consist of participants receiving on three consecutive days intramuscular (IM) injections of hydromorphone 0 mg (placebo), 6 mg and 18 mg doses during weeks 1-12 in randomized sequential order.
  Interventions: Drug: Buprenorphine; Drug: buprenorphine and naloxone; Drug: hydromorphone; Drug: placebo

INTERVENTIONS:
Drug: Buprenorphine — A subcutaneous depot injection of buprenorphine 300 mg was delivered using the ATRIGEL® Delivery System on study days 1 and 29. As the depot degrades, buprenorphine is released into systemic circulation over an extended period of time.
  Other Names: RBP-6000; Subcutaneous buprenorphine
Drug: buprenorphine and naloxone — Buprenorphine and naloxone (SUBOXONE® sublingual film) is given to participants on days -14 to day -1 (the SUBOXONE sublingual film stabilization period) or as soon as they start to experience withdrawal symptoms. SUBOXONE sublingual film may be initially administered several times daily until a stable dose between 8 mg and 24 mg daily is established.
  Other Names: SUBOXONE® sublingual film
Drug: hydromorphone — Hydromorphone IM challenges are administered during the screening period (days -17 to -15), on days -3 to -1 during the buprenorphine and naloxone (SUBOXONE sublingual film) stabilization period, and weekly during the 12-week treatment period after administration of RBP-6000. Each challenge consists of 3 days during which participants are randomly administered 0 mg (placebo), 6 mg and 18 mg hydromorphone via intramuscular (IM) injection daily in varying blinded sequences.
  Additionally, hydromorphone can also be earned during the afternoon Reinforcing effects tasks sessions up to the same randomized dose received in the hydromorphone challenge that morning (or money can be chosen).
  Other Names: dihydromorphinone
Drug: placebo — Placebo for hydromorphone administered via intramuscular injection during each challenge.
  Other Names: 0.45% normal saline

SUMMARY:
This is a multiple-dose study in non-treatment seeking male and female subjects with moderate to severe opioid use disorder who meet criteria from the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) to evaluate the effectiveness of RBP-6000 to block the effects of exogenous opioids.

The primary objective of this study was to demonstrate that the "Drug Liking" visual analog scale (VAS) measured after challenge with 6 mg (Dose 1) and 18 mg (Dose 2) hydromorphone was noninferior to the "Drug Liking" visual analog scale (VAS) measured after challenge with placebo at Weeks 1-4 post first injection of subcutaneous buprenorphine 300 mg (RBP-6000).

DETAILED DESCRIPTION:
For the hydromorphone challenge testing, subjects were randomized and assigned to 1 of 6 sequences during each week of hydromorphone challenge sessions.

On Day -18, subjects who met initial eligibility criteria were admitted to the clinical facility for the baseline hydromorphone challenge. If the subject had acceptable hydromorphone responses to the hydromorphone challenge, they remained confined to the clinical facility for induction on SUBOXONE sublingual film. Once it was confirmed that a subject was experiencing opioid withdrawal, as evidenced by a Clinical Opiate Withdrawal Scale (COWS) score greater than 12, the subject was inducted on SUBOXONE sublingual film. Multiple doses were allowed while subjects were reaching a stable dose until Day -9 when subjects were stabilized on a dose of SUBOXONE 8 mg - 24 mg. SUBOXONE sublingual film was administered daily at approximately the same time of day (± 1 hour) once the dose was stabilised. There was a hydromorphone challenge conducted on days -3 to -1. The last day of SUBOXONE dosing was day -1.

On Day 1, participants who met all inclusion/exclusion criteria and dosing criteria stopped receiving SUBOXONE sublingual film and received Injection 1 of RBP-6000 containing 300 mg buprenorphine. Participants returned in the evening of Days 4, 11, 18, and 25 to begin inpatient stays of 3 consecutive days (starting with Days 4-7 [and equivalent for subsequent weeks]). During these inpatient visits, subjects underwent randomised hydromorphone challenges, PK sample collection, Reinforcing Effects Tasks, and safety assessments.

On Day 29, participants received the second injection of RBP-6000 containing 300 mg buprenorphine (Injection 2). Participants returned in the evening on Days 32, 39, 46, 53, 60, 67, 74, and 81 to begin inpatient states of 3 consecutive days (starting with days 32-35 [and equivalent for subsequent weeks]). During these inpatient visits, subjects underwent randomised hydromorphone challenges, pharmacokinetic (PK) samples collection, Reinforcing Effects Tasks, and safety assessments. A window of ± 1 day was allowed for all visits, except the Day 53-56 visit, which was required by the protocol to be completed on those days.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for moderate or severe opioid use disorder at screening and are not seeking opioid use disorder treatment
* Body mass index of >= 18.0 to <= 33.0 kg/m^2
* Females - women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have negative pregnancy test prior to enrollment and must agree to use a medically acceptable means of contraception from screening through at least 3 months after the last dose of study drug
* Male subjects with female partners of child-bearing potential must agree to use medically acceptable contraception from screening through at least 3 months after the last dose of study drug

Exclusion Criteria:

* Subjects with any current diagnosis requiring chronic opioid treatment
* Subjects who currently meet the criteria for diagnosis of moderate or severe substance use disorder by DSM-5 criteria for any substances other than opioids, caffeine, or nicotine.
* Subjects who have abused or used buprenorphine within 14 days prior to informed consent.

Other protocol-defined criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Manager, Study Director — Indivior Inc.
Locations (1):
- Vince & Associates Clinical Research, Overland Park, Kansas, United States

REFERENCES:
- [Background] Greenwald MK, Johanson CE, Moody DE, Woods JH, Kilbourn MR, Koeppe RA, Schuster CR, Zubieta JK. Effects of buprenorphine maintenance dose on mu-opioid receptor availability, plasma concentrations, and antagonist blockade in heroin-dependent volunteers. Neuropsychopharmacology. 2003 Nov;28(11):2000-9. doi: 10.1038/sj.npp.1300251. PMID 12902992
- [Background] Greenwald M, Johanson CE, Bueller J, Chang Y, Moody DE, Kilbourn M, Koeppe R, Zubieta JK. Buprenorphine duration of action: mu-opioid receptor availability and pharmacokinetic and behavioral indices. Biol Psychiatry. 2007 Jan 1;61(1):101-10. doi: 10.1016/j.biopsych.2006.04.043. Epub 2006 Sep 1. PMID 16950210
- [Result] Nasser AF, Greenwald MK, Vince B, Fudala PJ, Twumasi-Ankrah P, Liu Y, Jones JP 3rd, Heidbreder C. Sustained-Release Buprenorphine (RBP-6000) Blocks the Effects of Opioid Challenge With Hydromorphone in Subjects With Opioid Use Disorder. J Clin Psychopharmacol. 2016 Feb;36(1):18-26. doi: 10.1097/JCP.0000000000000434. PMID 26650971
- [Derived] Laffont CM, Ngaimisi E, Gopalakrishnan M, Ivaturi V, Young M, Greenwald MK, Heidbreder C. Buprenorphine exposure levels to optimize treatment outcomes in opioid use disorder. Front Pharmacol. 2022 Nov 18;13:1052113. doi: 10.3389/fphar.2022.1052113. eCollection 2022. PMID 36467036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 342 subjects signed an informed consent with 39 subjects being enrolled and randomized to the sequential order of hydromorphone challenges to be received. The most common reason for not being randomized was due to the study exclusion criteria being met.
Groups:
- Depot Buprenorphine: Participants were treated with RBP-6000 300-mg in a single subcutaneous injection on Days 1 and 29. Challenges consist of participants receiving on three consecutive days intramuscular (IM) injections of hydromorphone randomly assigned at 0 mg (placebo), 6 mg and 18 mg doses during weeks 1-12.
Period: RBP-6000 Injection 1 (Day 1 to Day 28)
Arm/Group | Depot Buprenorphine
Started | 39
Intent to Treat Population | 38 (Subjects who receive >=1 dose of RBP-6000 and have >=1 complete sequence of hydromorphone challenges)
Completers Population | 30 (Subjects that reached Day 28 + completed all challenges at Week 4 were considered study completers.)
Completed | 30
Not Completed | 9
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 3
Period: RBP-6000 Injection 2 (Day 29 to Week 12)
Arm/Group | Depot Buprenorphine
Started | 30
Completed | 17
Not Completed | 13
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Depot Buprenorphine
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 79.55 (11.178)
Height [Mean (Standard Deviation); unit: cm] | 176.99 (6.421)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.35 (3.017)
Smoking History (Nicotine Use) [Mean (Standard Deviation); unit: years] — Population: 36 of 39 participants had a smoking history.
  years
    number analyzed (Participants) | 36
    (all) | 19.03 (8.962)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Blockade Following Administration of Hydromorphone Challenge As Measured Using the Subjective Opioid Effects Rating for the Question "Do You Like the Drug?" Visual Analog Scale (VAS) at Weeks 1-4 Analyzed by Mixed Model for Repeated Measures
Description: The study's primary objective was to determine if the opioid blocking effect for the first injection of buprenorphine 300 mg (RBP-6000) on Day 1 was not inferior to placebo when challenged by hydromorphone.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme liking of the drug 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone administration on the challenge days listed in the time frame field. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
Time Frame: Weeks 1 (Days 5-7), 2 (Days 12-14), 3 (Days 19-21), 4 (Days 26-28)
Population: The intent-to-treat (ITT) population included all subjects who received at least 1 dose of RBP-6000 and had at least 1 complete sequence (i.e., 0 mg [placebo], 6 mg and 18 mg hydromorphone in the randomised order) of hydromorphone challenges following administration of RBP-6000.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: During hydromorphone challenges, participants received intramuscular (IM) injections of placebo.
- Hydromorphone 6 mg: During hydromorphone challenges, participants received intramuscular (IM) injections of 6 mg hydromorphone.
- Hydromorphone 18 mg: During hydromorphone challenges, participants received intramuscular (IM) injections of 18 mg hydromorphone.
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Week 1 | 1.447 (1.638) | 5.103 (1.639) | 8.374 (1.638)
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 1.850 (1.216) | 2.436 (1.200) | 4.750 (1.200)
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.320 (1.476) | 2.183 (1.476) | 6.246 (1.475)
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.534 (2.214) | 3.849 (2.214) | 7.211 (2.214)
Statistical Analysis 1: Comparison: Placebo vs Hydromorphone 6 mg; Week 1 Complete hydromorphone blockade was claimed for RBP-6000 if blockade was achieved for both hydromorphone doses (6 mg and 18 mg) during each week of testing for the 4 weeks after the first dose of RBP-6000. Each test was performed at a 2-sided α = 0.05; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 3.656, 95% CI 2-sided [-0.032 to 7.344], Standard Error of Mean 1.850 — Hydromorphone - Placebo
Statistical Analysis 2: Comparison: Placebo vs Hydromorphone 18 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 6.927, 95% CI 2-sided [3.243 to 10.612], Standard Error of Mean 1.848 — Hydromorphone - Placebo
Statistical Analysis 3: Comparison: Placebo vs Hydromorphone 6 mg; Week 2 Complete hydromorphone blockade was claimed for RBP-6000 if blockade was achieved for both hydromorphone doses (6 mg and 18 mg) during each week of testing for the 4 weeks after the first dose of RBP-6000. Each test was performed at a 2-sided α = 0.05; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 0.586, 95% CI 2-sided [-1.977 to 3.149], Standard Error of Mean 1.283 — Hydromorphone - Placebo
Statistical Analysis 4: Comparison: Placebo vs Hydromorphone 18 mg; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 2.899, 95% CI 2-sided [0.333 to 5.465], Standard Error of Mean 1.285 — Hydromorphone - Placebo
Statistical Analysis 5: Comparison: Placebo vs Hydromorphone 6 mg; Week 3 Complete hydromorphone blockade was claimed for RBP-6000 if blockade was achieved for both hydromorphone doses (6 mg and 18 mg) during each week of testing for the 4 weeks after the first dose of RBP-6000. Each test was performed at a 2-sided α = 0.05; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 0.863, 95% CI 2-sided [-3.053 to 4.778], Standard Error of Mean 1.959 — Hydromorphone - Placebo
Statistical Analysis 6: Comparison: Placebo vs Hydromorphone 18 mg; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 4.926, 95% CI 2-sided [1.016 to 8.837], Standard Error of Mean 1.956 — Hydromorphone - Placebo
Statistical Analysis 7: Comparison: Placebo vs Hydromorphone 6 mg; Week 4 Complete hydromorphone blockade was claimed for RBP-6000 if blockade was achieved for both hydromorphone doses (6 mg and 18 mg) during each week of testing for the 4 weeks after the first dose of RBP-6000. Each test was performed at a 2-sided α = 0.05; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 3.316, 95% CI 2-sided [-1.425 to 8.025], Standard Error of Mean 2.367 — Hydromorphone - Placebo
Statistical Analysis 8: Comparison: Placebo vs Hydromorphone 18 mg; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority — Blockade was achieved if the upper bound of the 95% confidence interval was <= the non-inferiority margin of 11; LSM difference = 6.677, 95% CI 2-sided [1.936 to 11.418], Standard Error of Mean 2.367 — Hydromorphone - Placebo

2. Secondary Outcome: Reinforcing Effects (Breakpoint) by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Reinforcing Effects tasks began >= 5 hours after hydromorphone challenge. Participants made 12 choices between a preference for working for the amount of hydromorphone dosed that day or for money. The hydromorphone break point value is assigned to the highest level of hydromorphone units earned, with 1 unit having a breakpoint value of 5 and 12 units with a value of 2160.
  A repeated measures mixed-effects analysis of variance (ANOVA) was performed with the log transformed hydromorphone break point value as the dependent variable with period, hydromorphone sequence and hydromorphone dose as fixed effects, and subject nested within hydromorphone sequence as a random effect.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 4.984 [4.443 to 5.525] | 7.121 [6.746 to 7.497] | 7.042 [6.666 to 7.418]
  Week 1 | 4.767 [4.147 to 5.388] | 5.379 [4.784 to 5.975] | 5.708 [5.148 to 6.267]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 4.036 [3.229 to 4.842] | 4.779 [4.011 to 5.546] | 5.496 [4.835 to 6.157]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 4.760 [4.049 to 5.471] | 5.706 [5.024 to 6.388] | 5.669 [5.014 to 6.324]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 4.144 [3.382 to 4.907] | 5.533 [4.799 to 6.268] | 6.030 [5.326 to 6.733]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 4.564 [3.549 to 5.578] | 4.470 [3.517 to 5.424] | 4.936 [4.037 to 5.835]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 4.303 [3.210 to 5.396] | 4.419 [3.357 to 5.480] | 5.282 [4.291 to 6.273]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 5.092 [3.745 to 6.440] | 5.808 [4.455 to 7.161] | 5.965 [4.628 to 7.303]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 3.899 [2.780 to 5.019] | 4.418 [3.341 to 5.494] | 4.747 [3.646 to 5.849]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 4.342 [3.116 to 5.568] | 4.432 [3.383 to 5.481] | 5.437 [4.506 to 6.368]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 4.546 [2.970 to 6.122] | 4.578 [2.995 to 6.161] | 4.997 [3.444 to 6.551]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 4.330 [2.958 to 5.702] | 4.114 [2.865 to 5.364] | 5.076 [3.906 to 6.247]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 4.029 [3.151 to 4.906] | 4.623 [3.588 to 5.659] | 5.615 [4.726 to 6.503]

3. Secondary Outcome: Reinforcing Effects Of the Daily Randomized Hydromorphone Challenge as Measured by the Mean Hydromorphone Break Point Value at Weeks 1-12
Description: The ability of RBP-6000 to reduce the reinforcing effects of hydromorphone used money as a choice alternative to hydromorphone.
  Reinforcing Effects Tasks began no earlier than 5 hours after randomised hydromorphone administration for each day. Each test consisted of the participant making 12 choices between a preference for working for the amount of hydromorphone dosed earlier that day or for money (each choice therefore has a scale of 0-12). The hydromorphone break point value is the ratio of the highest number of choices for hydromorphone to the highest number of choices for money. Hydromorphone breakpoint values were then analysed by week using a repeated measures mixed-effects model with period, hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect. Analyses were carried out on the log10 transformed hydromorphone breakpoint value.
Time Frame: Weeks 1 (Days 5-7), 2 (Days 12-14), 3 (Days 19-21), 4 (Days 26-28), 5 (Days 33-35), 6 (Days 40-42), 7 (Days 47-49), 8 (Days 53-56), 9 (Days 61-63), 10 (Days 68-70), 11 (Days 75-77), 12 (Days 82-84)
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: log10 transformed ratio
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
log10 transformed ratio
  Week 1 | 2.070 (0.134) | 2.336 (0.129) | 2.479 (0.120)
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 1.753 (0.175) | 2.075 (0.166) | 2.387 (0.142)
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 2.067 (0.153) | 2.478 (0.146) | 2.462 (0.140)
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 1.800 (0.164) | 2.403 (0.158) | 2.619 (0.151)
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 1.982 (0.217) | 1.941 (0.203) | 2.144 (0.190)
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 1.869 (0.232) | 1.919 (9.224) | 2.294 (0.208)
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 2.212 (0.277) | 2.522 (0.278) | 2.591 (0.274)
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 1.694 (0.232) | 1.919 (0.220) | 2.062 (0.227)
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 1.886 (0.262) | 1.925 (0.224) | 2.361 (0.197)
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 1.974 (0.310) | 1.988 (0.313) | 2.170 (0.302)
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 1.880 (0.289) | 1.787 (0.261) | 2.205 (0.242)
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 1.750 (0.180) | 2.008 (0.217) | 2.438 (0.183)

4. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: TEAE=any untoward medical occurrence that develops or worsens in severity after administration of study drug and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= a marked limitation in activity. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required intervention to prevent one of the outcomes listed above.
  All adverse events that occurred between Day 1 to Day 91 are reported under the Depot Buprenorphine treatment arm.
  Adverse events that occurred on the day of a hydromorphone challenge are also reported under the appropriate hydromorphone challenge arm.
Time Frame: Depot Buprenorphine: Day 1 to Day 91. The three hydromorphone challenge levels were randomly assigned to one day in each of the three-day groupings spanning 12 weeks: Days 5-7, 11-14, 19-21, 26-28, 33-35, 40-42, 47-49, 54-56, 61-63, 68-70, 75-77, 82-84
Population: Safety; one participant was administered the first RBP-6000 injection but no hydromorphone challenges. Investigators did not assess AEs for potential relatedness to hydromorphone.
Measure: Count of Participants; unit: Participants
Groups:
- Depot Buprenorphine: Participants were treated with RBP-6000 300-mg in a single subcutaneous injection on Days 1 and 29.
- Placebo Challenge: Participants received three hydromorphone challenges each week, one challenge on each of three consecutive days/week in this 12 week study. Participants and clinical facility staff were blinded to the specific dose of hydromorphone being administered during each challenge.
  The placebo challenge consisted of an intramuscular injection of placebo (hydromorphone 0mg).
- Hydromorphone 6 mg Challenge: Participants received three hydromorphone challenges each week, one challenge on each of three consecutive days/week in this 12 week study. Participants and clinical facility staff were blinded to the specific dose of hydromorphone being administered during each challenge.
  The hydromorphone 6 mg challenge consisted of an intramuscular injection of 6 mg hydromorphone.
- Hydromorphone 18 mg Challenge: Participants received three hydromorphone challenges each week, one challenge on each of three consecutive days/week in this 12 week study. Participants and clinical facility staff were blinded to the specific dose of hydromorphone being administered during each challenge.
  The hydromorphone 18 mg challenge consisted of an intramuscular injection of 18 mg hydromorphone.
Arm/Group | Depot Buprenorphine | Placebo Challenge | Hydromorphone 6 mg Challenge | Hydromorphone 18 mg Challenge
Number analyzed (Participants) | 39 | 38 | 38 | 38
Participants
  >=1 TEAE | 39 | 29 | 26 | 25
  >=1 TEAE related to study drug: number analyzed (Participants) | 39 | 0 | 0 | 0
  >=1 TEAE related to study drug | 25 |  |  |
  >=1 Severe TEAE | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0
  >=1 SAE other than death | 0 | 0 | 0 | 0
  Withdrew from study due to a TEAE | 0 | 0 | 0 | 0

5. Secondary Outcome: Plasma Concentrations of Buprenorphine Summarized by Study Week
Description: PK Sampling Schedule:
  * Day -17 to -15: before hydromorphone admin
  * Day -4: before Suboxone admin
  * Day 2: 24 hours after RBP-6000 admin
  * Days 5-7, 12-14, 19-21 and 26-28: immediately before hydromorphone admin
  * Days 29: before RBP-6000 admin
  * Day 30: 24 hours after RBP-6000 admin
  * Days 33-35, 40-42, 47-49, 54-56, 61-63, 68-70, 75-77, and 82-84: immediately before hydromorphone admin
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
ng/mL
  Week -1 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Week 1 | 2.030 (0.717) | 2.164 (0.882) | 2.042 (0.765)
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 1.892 (0.637) | 1.874 (0.605) | 1.970 (0.764)
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.933 (0.657) | 1.882 (0.663) | 1.916 (0.606)
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 1.722 (0.648) | 1.776 (0.602) | 1.812 (0.633)
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 3.684 (1.174) | 3.649 (1.122) | 3.667 (1.035)
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 3.423 (1.082) | 3.530 (1.104) | 3.521 (1.181)
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 3.427 (1.121) | 3.495 (1.107) | 3.466 (1.136)
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 3.326 (1.217) | 3.365 (1.160) | 3.497 (1.304)
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 3.156 (1.103) | 3.122 (1.030) | 3.210 (1.200)
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 2.985 (1.074) | 3.039 (3.193) | 1.150 (1.136)
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 3.117 (1.257) | 2.985 (3.081) | 1.083 (1.124)
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 2.626 (0.956) | 2.646 (1.039) | 2.624 (0.945)

6. Secondary Outcome: Predicted mu Opioid Receptor Occupancy (μORO) by Mean Buprenorphine Concentrations and Study Week
Description: A population pharmacokinetic/pharmacodynamic (PK/PD) model was developed to model the relationship between buprenorphine plasma concentrations and brain μORO based on 2 published clinical trials. This model used individual buprenorphine plasma concentrations measured to derive muORO individual predictions that were further described using summary statistics. The relationship between buprenorphine plasma concentration and μORO was best described by a maximal effect (Emax) model:
  µORO = E(max)*Cp / EC(50) + Cp
  Where Cp is the plasma concentration of buprenorphine, Emax is the maximal μORO, and EC50 is the plasma concentration of buprenorphine that is expected to achieve 50% of the maximal μORO. A direct (instantaneous) relationship between buprenorphine plasma concentration and µORO, i.e. without equilibration delay, was assumed.
  Row title format: Study Week: buprenorphine plasma concentrations for placebo/ 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population
Measure: Mean (Standard Deviation); unit: percentage receptor occupancy
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
percentage receptor occupancy
  Baseline Week -1: 0.00/0.00/0.00 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Week 1: 2.03/2.16/2.04 | 67.077 (6.675) | 67.875 (6.806) | 67.089 (6.591)
  Week 2: 1.89/1.87/1.97: number analyzed (Participants) | 34 | 35 | 35
  Week 2: 1.89/1.87/1.97 | 66.071 (6.240) | 66.059 (5.692) | 66.485 (6.670)
  Week 3: 1.93/1.88/1.92: number analyzed (Participants) | 33 | 33 | 33
  Week 3: 1.93/1.88/1.92 | 66.442 (6.108) | 66.000 (6.010) | 66.438 (5.934)
  Week 4: 1.72/1.78/1.81: number analyzed (Participants) | 30 | 30 | 30
  Week 4: 1.72/1.78/1.81 | 64.270 (6.116) | 65.108 (5.534) | 65.349 (5.848)
  Week 5: 3.68/3.65/3.67: number analyzed (Participants) | 29 | 28 | 30
  Week 5: 3.68/3.65/3.67 | 76.346 (4.031) | 76.285 (3.938) | 76.417 (3.856)
  Week 6: 3.42/3.53/3.52: number analyzed (Participants) | 27 | 27 | 27
  Week 6: 3.42/3.53/3.52 | 75.432 (4.156) | 75.699 (4.685) | 75.686 (4.366)
  Week 7: 3.43/3.50/3.47: number analyzed (Participants) | 27 | 26 | 27
  Week 7: 3.43/3.50/3.47 | 75.351 (4.347) | 75.641 (4.373) | 75.429 (4.601)
  Week 8: 3.33/3.37/3.50: number analyzed (Participants) | 24 | 24 | 24
  Week 8: 3.33/3.37/3.50 | 74.544 (5.419) | 74.792 (5.495) | 75.179 (5.302)
  Week 9: 3.16/3.12/3.21: number analyzed (Participants) | 22 | 22 | 22
  Week 9: 3.16/3.12/3.21 | 74.000 (5.314) | 73.970 (5.131) | 74.036 (5.692)
  Week 10: 2.99/3.04/3.19: number analyzed (Participants) | 20 | 19 | 19
  Week 10: 2.99/3.04/3.19 | 73.002 (6.288) | 73.075 (6.579) | 74.179 (5.355)
  Week 11: 3.12/2.99/3.08: number analyzed (Participants) | 18 | 18 | 18
  Week 11: 3.12/2.99/3.08 | 73.385 (6.382) | 73.054 (6.099) | 73.507 (5.904)
  Week 12: 2.63/2.65/2.62: number analyzed (Participants) | 17 | 17 | 17
  Week 12: 2.63/2.65/2.62 | 71.274 (5.946) | 71.313 (5.933) | 71.303 (5.863)

7. Secondary Outcome: Change From Placebo in Reinforcing Effects (Breakpoint) by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: This endpoint explores the correlation between the reinforcing effects of hydromorphone and simulated mu opioid receptor occupancy.
  Data are reported as change from placebo least square mean of Log10 transformed values for reinforcing effects. Reinforcing Effects tasks began >= 5 hours after hydromorphone challenge. Participants made 12 choices between a preference for working for the amount of hydromorphone dosed that day or for money. The hydromorphone break point value is assigned to the highest level of hydromorphone units earned, with 1 unit having a breakpoint value of 5 and 12 units with a value of 2160.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: predicted mu opioid receptor occupancy for 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 transformed ratio
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
log10 transformed ratio
  Baseline Week -1: 0.00/0.00 % | 0.93 [0.67 to 1.18] | 0.89 [0.64 to 1.17]
  Week 1: 67.88/67.09 % | 0.27 [-0.001 to 0.53] | 0.41 [0.15 to 0.67]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 0.32 [-0.05 to 0.70] | 0.63 [0.28 to 0.99]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 0.41 [0.14 to 0.69] | 0.40 [0.13 to 0.66]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | 0.60 [0.31 to 0.90] | 0.82 [0.53 to 1.11]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | -0.04 [-0.47 to 0.39] | 0.16 [-0.24 to 0.56]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | 0.05 [-0.41 to 0.51] | 0.43 [-0.03 to 0.88]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | 0.31 [-0.004 to 0.63] | 0.38 [0.043 to 0.72]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | 0.23 [-0.16 to 0.61] | 0.37 [-0.05 to 0.79]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | 0.04 [-0.61 to 0.69] | 0.48 [-0.14 to 1.09]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | 0.01 [-0.41 to 0.44] | 0.20 [-0.22 to 0.61]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | -0.09 [-0.73 to 0.55] | 0.32 [-0.29 to 0.94]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | 0.26 [-0.25 to 0.77] | 0.69 [0.22 to 1.16]

8. Secondary Outcome: Visual Analog Scale (VAS) Score for "Do You Like the Drug?" by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme liking of the drug 30 minutes before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 2.892 [-5.079 to 10.862] | 48.252 [40.223 to 56.281] | 63.503 [55.443 to 71.562]
  Week 1 | 1.447 [-1.813 to 4.707] | 5.103 [1.840 to 8.366] | 8.374 [5.113 to 11.636]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 1.850 [-0.578 to 4.279] | 2.436 [0.038 to 4.835] | 4.750 [2.351 to 7.148]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.320 [-1.615 to 4.255] | 2.183 [-0.752 to 5.118] | 6.246 [3.314 to 9.179]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.534 [-3.906 to 4.973] | 3.849 [-0.590 to 8.289] | 7.211 [2.771 to 11.650]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 1.048 [-0.495 to 2.590] | 1.785 [0.220 to 3.349] | 2.258 [0.733 to 3.783]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 0.440 [-2.495 to 3.375] | 0.789 [-2.146 to 3.723] | 3.600 [0.68 to 6.542]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 0.672 [-0.839 to 2.183] | 0.521 [-1.021 to 2.063] | 2.550 [1.040 to 4.061]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 1.270 [-2.052 to 4.592] | 0.225 [-3.090 to 3.540] | 3.203 [-0.112 to 6.518]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 0.451 [-3.982 to 4.884] | 0.328 [-4.122 to 4.777] | 4.616 [0.200 to 9.032]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 0.596 [-0.153 to 1.345] | 0.507 [-0.253 to 1.268] | 0.722 [-0.041 to 1.485]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 1.471 [-1.135 to 4.076] | 1.154 [-1.451 to 3.760] | 4.709 [2.135 to 7.283]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 0.973 [-0.644 to 2.589] | 0.939 [-0.722 to 2.599] | 3.756 [2.085 to 5.427]

9. Secondary Outcome: Change From Placebo in VAS Score for "Do You Like the Drug?" by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme liking of the drug 30 minutes before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo. For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: mean predicted mu opioid receptor occupancy for 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Week -1: 0.00/0.00 % | 45.36 [37.16 to 53.56] | 60.61 [52.32 to 68.90]
  Week 1: 67.88/67.09 % | 3.66 [-0.03 to 7.34] | 6.93 [3.24 to 10.61]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 0.59 [-1.98 to 3.15] | 2.90 [0.33 to 5.47]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 0.86 [-3.05 to 4.78] | 4.93 [1.02 to 8.84]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | 3.32 [-1.43 to 8.06] | 6.68 [1.94 to 11.42]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | 0.74 [-0.94 to 2.42] | 1.21 [-0.43 to 2.85]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | 0.35 [-3.62 to 4.32] | 3.16 [-0.83 to 7.15]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | -0.15 [-2.16 to 1.86] | 1.88 [-0.11 to 3.87]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | -1.05 [-4.77 to 2.68] | 1.93 [-1.79 to 5.66]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | -0.12 [-6.20 to 5.96] | 4.17 [-1.84 to 10.17]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | -0.09 [-0.69 to 0.51] | 0.13 [-0.50 to 0.76]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | -0.32 [-3.97 to 3.34] | 3.24 [-0.35 to 6.83]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | -0.03 [-2.19 to 2.12] | 2.78 [0.61 to 4.96]

10. Secondary Outcome: VAS Score for "How High Are You Right Now?" by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme high from the drug 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 2.654 [-4.624 to 9.932] | 33.052 [25.722 to 40.382] | 53.597 [46.239 to 60.954]
  Week 1 | 1.386 [-1.261 to 4.034] | 4.444 [1.795 to 7.093] | 6.240 [3.592 to 8.889]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 2.020 [-0.639 to 4.679] | 2.539 [-0.089 to 5.167] | 5.173 [2.545 to 7.801]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.362 [-1.380 to 4.103] | 3.028 [0.286 to 5.769] | 5.731 [2.991 to 8.471]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.595 [-3.818 to 5.007] | 4.251 [-0.161 to 8.663] | 7.737 [3.325 to 12.149]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 0.860 [-0.800 to 2.521] | 2.406 [0.726 to 4.085] | 2.304 [0.660 to 3.948]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 0.463 [-1.426 to 2.351] | 0.878 [-1.010 to 2.767] | 2.555 [0.662 to 4.448]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 0.661 [-0.777 to 2.099] | 0.540 [-0.927 to 2.008] | 2.481 [1.043 to 3.919]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 1.431 [-1.947 to 4.810] | 0.261 [-3.111 to 3.633] | 3.277 [-0.095 to 6.649]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 0.519 [-3.869 to 4.906] | 0.265 [-4.139 to 4.669] | 4.534 [0.163 to 8.905]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 0.644 [0.011 to 1.277] | 0.417 [-0.221 to 1.056] | 0.624 [-0.016 to 1.263]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 0.950 [0.023 to 1.877] | 0.987 [0.060 to 1.914] | 2.460 [1.540 to 3.379]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 0.289 [-0.847 to 1.426] | 0.458 [-0.680 to 1.597] | 0.994 [-0.145 to 2.133]

11. Secondary Outcome: Change From Placebo in VAS Score for "How High Are You Right Now?" by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme high from the drug 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo. For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: mean predicted mu opioid receptor occupancy 6 mg / 18 mg
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Week -1: 0.00/0.00 % | 30.40 [22.99 to 37.81] | 50.94 [43.45 to 58.43]
  Week 1: 67.88/67.09 % | 3.06 [0.35 to 5.76] | 4.85 [2.15 to 7.56]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 0.52 [-2.20 to 3.23] | 3.15 [0.44 to 5.87]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 1.67 [-1.78 to 5.11] | 4.37 [0.93 to 7.81]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | 3.66 [-1.21 to 8.52] | 7.14 [2.28 to 12.01]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | 1.55 [-0.08 to 3.18] | 1.44 [-0.15 to 3.03]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | 0.42 [-2.01 to 2.84] | 2.09 [-0.35 to 4.53]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | -0.12 [-2.01 to 1.77] | 1.82 [-0.05 to 3.69]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | -1.17 [-4.88 to 2.54] | 1.85 [-1.87 to 5.56]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | -0.25 [-6.29 to 5.78] | 4.02 [-1.94 to 9.97]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | -0.23 [-0.60 to 0.14] | -0.02 [-0.41 to 0.37]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | 0.04 [-1.07 to 1.14] | 1.51 [0.43 to 2.59]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | 0.17 [-0.29 to 0.63] | 0.71 [0.24 to 1.17]

12. Secondary Outcome: VAS Score for "Do You Feel Any Drug Effect?" by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme drug effect 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 3.274 [-3.844 to 10.391] | 39.047 [31.880 to 46.213] | 58.912 [51.720 to 66.105]
  Week 1 | 1.200 [-1.172 to 3.572] | 4.214 [1.840 to 6.588] | 6.433 [4.060 to 8.806]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 1.775 [-0.751 to 4.302] | 2.787 [0.290 to 5.284] | 5.466 [2.969 to 7.962]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.193 [-1.605 to 3.992] | 2.933 [0.135 to 5.732] | 6.046 [3.249 to 8.842]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.514 [-4.058 to 5.086] | 4.491 [-0.081 to 9.063] | 8.269 [3.697 to 12.841]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 0.933 [-0.798 to 2.665] | 2.497 [0.746 to 4.247] | 2.388 [0.673 to 4.103]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 0.673 [-0.154 to 1.500] | 0.872 [0.045 to 1.699] | 1.364 [0.536 to 2.191]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 0.625 [-0.688 to 1.939] | 0.533 [-0.808 to 1.874] | 2.269 [0.955 to 3.583]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 1.297 [-2.011 to 4.604] | 0.329 [-2.971 to 3.630] | 3.240 [-0.061 to 6.540]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 0.522 [-3.864 to 4.907] | 0.305 [-4.098 to 4.708] | 5.033 [0.665 to 9.402]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 0.654 [-0.083 to 1.390] | 0.491 [-0.256 to 1.238] | 0.709 [-0.040 to 1.457]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 0.993 [-0.050 to 2.037] | 1.118 [0.074 to 2.162] | 2.935 [1.903 to 3.966]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 0.285 [-0.809 to 1.379] | 0.524 [-0.573 to 1.621] | 1.269 [0.172 to 2.367]

13. Secondary Outcome: Change From Placebo in VAS Score for "Do You Feel Any Drug Effect?" by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme drug effect 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo. For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: mean predicted mu opioid receptor occupancy for 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Week -1: 0.00/0.00 % | 35.77 [28.66 to 42.89] | 55.64 [48.45 to 62.83]
  Week 1: 67.88/67.09 % | 3.01 [0.44 to 5.58] | 5.23 [2.67 to 7.80]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 1.01 [-1.60 to 3.62] | 3.69 [1.08 to 6.30]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 1.74 [-1.75 to 5.23] | 4.85 [1.37 to 8.34]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | 3.98 [-1.01 to 8.97] | 7.76 [2.77 to 12.74]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | 1.56 [-0.09 to 3.22] | 1.46 [-0.16 to 3.07]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | 0.20 [-0.70 to 1.10] | 0.69 [-0.21 to 1.59]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | -0.09 [-1.82 to 1.64] | 1.64 [-0.07 to 3.35]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | -0.97 [-4.70 to 2.76] | 1.94 [-1.79 to 5.67]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | -0.22 [-6.32 to 5.89] | 4.51 [-1.52 to 10.54]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | -0.16 [-0.71 to 0.39] | 0.06 [-0.52 to 0.63]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | 0.13 [-1.34 to 1.59] | 1.94 [0.50 to 3.38]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | 0.24 [-0.28 to 0.76] | 0.98 [0.46 to 1.51]

14. Secondary Outcome: VAS Score for "Does the Drug Have Any Good Effects?" by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme good effect 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 3.131 [-4.201 to 10.464] | 43.888 [36.500 to 51.276] | 61.640 [54.223 to 69.057]
  Week 1 | 1.239 [-1.658 to 4.135] | 4.252 [1.352 to 7.151] | 7.072 [4.174 to 9.970]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 1.768 [-0.820 to 4.356] | 2.364 [-0.193 to 4.922] | 5.263 [2.706 to 7.821]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.221 [-2.599 to 5.041] | 2.930 [-0.890 to 6.750] | 7.395 [3.578 to 11.212]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.476 [-4.098 to 5.050] | 4.508 [-0.066 to 9.082] | 8.130 [3.556 to 12.704]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 0.863 [-0.813 to 2.538] | 2.264 [0.569 to 3.959] | 2.270 [0.612 to 3.929]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 0.410 [-0.377 to 1.197] | 0.761 [-0.026 to 1.548] | 1.164 [0.376 to 1.952]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 0.574 [-0.755 to 1.902] | 0.504 [-0.852 to 1.861] | 2.225 [0.896 to 3.554]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 1.289 [-2.063 to 4.641] | 0.188 [-3.157 to 3.533] | 3.146 [-0.199 to 6.491]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 0.399 [-4.028 to 4.825] | 0.270 [-4.173 to 4.714] | 4.815 [0.405 to 9.225]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 0.536 [-0.155 to 1.226] | 0.564 [-0.137 to 1.265] | 0.681 [-0.022 to 1.384]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 1.149 [-0.679 to 2.978] | 1.023 [-0.805 to 2.851] | 3.712 [1.906 to 5.518]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 0.550 [-0.616 to 1.716] | 0.681 [-0.498 to 1.860] | 2.251 [1.069 to 3.433]

15. Secondary Outcome: Change From Placebo in VAS Score for "Does the Drug Have Any Good Effects?" by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme good effect 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo. For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: mean predicted mu opioid receptor occupancy for 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Week -1: 0.00/0.00 % | 40.76 [33.10 to 48.42] | 58.51 [50.76 to 66.26]
  Week 1: 67.88/67.09 % | 3.01 [-0.28 to 6.30] | 5.83 [2.55 to 9.12]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 0.60 [-2.08 to 3.27] | 3.50 [0.82 to 6.17]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 1.71 [-3.36 to 6.78] | 6.17 [1.11 to 11.24]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | 4.03 [-0.82 to 8.88] | 7.65 [2.81 to 12.50]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | 1.40 [-0.27 to 3.07] | 1.41 [-0.22 to 3.03]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | 0.35 [-0.45 to 1.15] | 0.75 [-0.05 to 1.55]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | -0.07 [-1.84 to 1.70] | 1.65 [-0.10 to 3.40]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | -1.10 [-4.86 to 2.66] | 1.86 [-1.90 to 5.62]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | -0.13 [-6.23 to 5.98] | 4.42 [-1.61 to 10.45]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | 0.03 [-0.51 to 0.57] | 0.15 [-0.42 to 0.71]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | -0.13 [-2.69 to 2.44] | 2.56 [0.04 to 5.08]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | 0.13 [-0.96 to 1.22] | 1.70 [0.60 to 2.80]

16. Secondary Outcome: VAS Score for "Does the Drug Have Any Bad Effects?" by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme bad effect 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 4.797 [0.690 to 8.904] | 7.145 [3.027 to 11.262] | 11.046 [6.909 to 15.183]
  Week 1 | 1.117 [0.595 to 1.638] | 1.159 [0.638 to 1.681] | 1.107 [0.586 to 1.629]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 0.980 [0.282 to 1.677] | 1.120 [0.430 to 1.810] | 1.507 [0.817 to 2.197]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 0.842 [0.237 to 1.447] | 0.926 [0.321 to 1.531] | 1.228 [0.623 to 1.833]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.691 [0.146 to 1.235] | 0.663 [0.118 to 1.208] | 1.117 [0.572 to 1.662]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 0.785 [0.450 to 1.119] | 0.817 [0.481 to 1.152] | 0.690 [0.356 to 1.024]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 0.494 [0.116 to 0.872] | 0.521 [0.143 to 0.899] | 0.525 [0.147 to 0.903]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 0.760 [0.411 to 1.110] | 0.666 [0.316 to 1.016] | 0.642 [0.292 to 0.992]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 0.544 [0.101 to 0.987] | 0.553 [0.110 to 0.996] | 0.508 [0.065 to 0.951]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 0.376 [-0.088 to 0.839] | 0.395 [-0.068 to 0.858] | 0.434 [-0.029 to 0.897]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 0.504 [-0.037 to 1.046] | 0.420 [-0.122 to 0.962] | 0.403 [-0.139 to 0.945]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 0.523 [-0.006 to 1.051] | 0.629 [0.101 to 1.157] | 0.569 [0.041 to 1.097]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 0.393 [-0.415 to 1.201] | 0.387 [-0.421 to 1.195] | 0.368 [-0.440 to 1.176]

17. Secondary Outcome: Change From Placebo in VAS Score for "Does the Drug Have Any Bad Effects?" by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme bad effect 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo. For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: mean predicted mu opioid receptor occupancy for 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Week -1: 0.00/0.00 % | 2.35 [-1.19 to 5.88] | 6.25 [2.64 to 9.85]
  Week 1: 67.88/67.09 % | 0.04 [-0.16 to 0.25] | -0.01 [-0.21 to 0.19]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 0.14 [-0.55 to 0.83] | 0.53 [-0.16 to 1.22]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 0.08 [-0.54 to 0.71] | 0.39 [-0.24 to 1.01]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | -0.03 [-0.52 to 0.47] | 0.43 [-0.07 to 0.92]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | 0.03 [-0.13 to 0.19] | -0.10 [-0.25 to 0.06]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | 0.03 [-0.14 to 0.20] | 0.03 [-0.14 to 0.20]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | -0.09 [-0.25 to 0.06] | -0.12 [-0.27 to 0.03]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | 0.01 [-0.11 to 0.13] | -0.04 [-0.16 to 0.09]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | 0.02 [-0.08 to 0.12] | 0.06 [-0.04 to 0.16]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | -0.08 [-0.20 to 0.03] | -0.10 [-0.22 to 0.02]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | 0.11 [-0.04 to 0.25] | 0.05 [-0.10 to 0.19]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | -0.01 [-0.11 to 0.10] | -0.02 [-0.13 to 0.08]

18. Secondary Outcome: VAS Score for "Do You Feel Sedated?" by Study Week Analyzed by Mixed Model for Repeated Measures
Description: This outcome reports observed values used in the "Change from Placebo....' endpoint that follows.
  Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme sedation 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo.
  For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Blockade is achieved if the upper bound of the 95% confidence interval is <= to the non-inferiority margin of 11.
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38 | 38
units on a scale
  Baseline Week -1 | 3.399 [-3.436 to 10.235] | 14.504 [7.640 to 21.367] | 30.979 [24.068 to 37.890]
  Week 1 | 1.199 [-1.859 to 4.256] | 3.979 [0.920 to 7.038] | 5.401 [2.344 to 8.457]
  Week 2: number analyzed (Participants) | 34 | 35 | 35
  Week 2 | 3.126 [-0.702 to 6.954] | 3.508 [-0.296 to 7.312] | 7.048 [3.245 to 10.852]
  Week 3: number analyzed (Participants) | 33 | 33 | 33
  Week 3 | 1.135 [-1.565 to 3.835] | 1.975 [-0.725 to 4.675] | 4.897 [2.199 to 7.594]
  Week 4: number analyzed (Participants) | 30 | 30 | 30
  Week 4 | 0.661 [-3.518 to 4.839] | 3.462 [-0.717 to 7.640] | 5.774 [1.596 to 9.952]
  Week 5: number analyzed (Participants) | 29 | 28 | 30
  Week 5 | 1.110 [-1.150 to 3.369] | 2.873 [0.588 to 5.158] | 2.445 [0.207 to 4.682]
  Week 6: number analyzed (Participants) | 27 | 27 | 27
  Week 6 | 1.152 [-1.488 to 3.793] | 0.923 [-1.718 to 3.563] | 3.354 [0.708 to 6.000]
  Week 7: number analyzed (Participants) | 27 | 26 | 27
  Week 7 | 2.348 [-1.871 to 6.567] | 2.233 [-2.001 to 6.468] | 3.894 [-0.325 to 8.113]
  Week 8: number analyzed (Participants) | 24 | 24 | 24
  Week 8 | 1.787 [-2.647 to 6.220] | 1.142 [-3.286 to 5.571] | 3.395 [-1.033 to 7.824]
  Week 9: number analyzed (Participants) | 22 | 22 | 22
  Week 9 | 0.506 [-4.077 to 5.088] | 1.041 [-3.557 to 5.639] | 4.996 [0.429 to 9.564]
  Week 10: number analyzed (Participants) | 20 | 19 | 19
  Week 10 | 1.155 [-0.144 to 2.454] | 0.567 [-0.766 to 1.900] | 1.032 [-0.312 to 2.375]
  Week 11: number analyzed (Participants) | 18 | 18 | 18
  Week 11 | 0.858 [-1.372 to 3.088] | 1.403 [-0.827 to 3.633] | 3.299 [1.085 to 5.512]
  Week 12: number analyzed (Participants) | 17 | 17 | 17
  Week 12 | 0.344 [-2.035 to 2.723] | 2.408 [-0.024 to 4.841] | 0.086 [-2.360 to 2.532]

19. Secondary Outcome: Change From Placebo in VAS Score for "Do You Feel Sedated?" by Study Week and Simulated mu Opioid Receptor Occupancy (μORO)
Description: Participants completed a visual analog scale (VAS) that ranged from 0 - 100, with 0 meaning not at all, and 100 meaning the most extreme sedation 30 minutes (± 5 minutes) before and 15, 30 , 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, and 300 minutes (± 5 minutes) after hydromorphone challenge. The drug in question was hydromorphone (6 or 18 mg) or placebo. For each hydromorphone challenge week, a mixed-effects model with period (where period is day), hydromorphone sequence, and hydromorphone dose as fixed effects and subject nested within hydromorphone sequence as a random effect were used for analysis.
  Change from placebo was calculated as Active Challenge result - Placebo Challenge result. Values that approach 0 (implying little difference between the Active Challenge result and the Placebo Challenge result) indicate effectiveness of the opioid blockade.
  Row titles include Study Week: mean predicted mu opioid receptor occupancy for 6 mg / 18 mg challenge dosages
Time Frame: Baseline (Week -1), Weeks 1-12 (RBP-6000 admin on Weeks 1 and 5)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hydromorphone 6 mg | Hydromorphone 18 mg
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Week -1: 0.00/0.00 % | 11.10 [3.99 to 18.22] | 27.58 [20.32 to 34.84]
  Week 1: 67.88/67.09 % | 2.78 [-0.001 to 5.56] | 4.20 [1.43 to 6.97]
  Week 2: 66.06/66.49 %: number analyzed (Participants) | 35 | 35
  Week 2: 66.06/66.49 % | 0.38 [-2.52 to 3.28] | 3.92 [1.02 to 6.83]
  Week 3: 66.00/66.44 %: number analyzed (Participants) | 33 | 33
  Week 3: 66.00/66.44 % | 0.84 [-2.71 to 4.39] | 3.76 [0.22 to 7.31]
  Week 4: 65.11/65.35 %: number analyzed (Participants) | 30 | 30
  Week 4: 65.11/65.35 % | 2.80 [-1.54 to 7.14] | 5.11 [0.78 to 9.45]
  Week 5: 76.29/76.42 %: number analyzed (Participants) | 28 | 30
  Week 5: 76.29/76.42 % | 1.76 [-0.44 to 3.97] | 1.34 [-0.82 to 3.49]
  Week 6: 75.70/75.69 %: number analyzed (Participants) | 27 | 27
  Week 6: 75.70/75.69 % | -0.23 [-3.59 to 3.13] | 2.20 [-1.17 to 5.58]
  Week 7: 75.64/75.43 %: number analyzed (Participants) | 26 | 27
  Week 7: 75.64/75.43 % | -0.12 [-2.35 to 2.12] | 1.55 [-0.66 to 3.75]
  Week 8: 74.79/75.18 %: number analyzed (Participants) | 24 | 24
  Week 8: 74.79/75.18 % | -0.64 [-4.51 to 3.22] | 1.61 [-2.26 to 5.47]
  Week 9: 73.97/74.04 %: number analyzed (Participants) | 22 | 22
  Week 9: 73.97/74.04 % | 0.54 [-5.39 to 6.46] | 4.49 [-1.36 to 10.34]
  Week 10: 73.08/74.18 %: number analyzed (Participants) | 19 | 19
  Week 10: 73.08/74.18 % | -0.59 [-2.01 to 0.84] | -0.12 [-1.61 to 1.36]
  Week 11: 73.05/73.51 %: number analyzed (Participants) | 18 | 18
  Week 11: 73.05/73.51 % | 0.55 [-2.00 to 3.10] | 2.44 [-0.06 to 4.94]
  Week 12: 71.31/71.30 %: number analyzed (Participants) | 17 | 17
  Week 12: 71.31/71.30 % | 2.06 [-0.93 to 5.06] | -0.26 [-3.29 to 2.77]

ADVERSE EVENTS:
Time Frame: Depot Buprenorphine: Day 1 to Day 91. Hydromorphone Challenges: the three hydromorphone challenge levels (0 mg, 6 mg and 18 mg) were randomly assigned to one day in each of the three-day groupings spanning 12 weeks: Days 5-7, 11-14, 19-21, 26-28, 33-35, 40-42, 47-49, 54-56, 61-63, 68-70, 75-77, and 82-84.
Description: All adverse events that occurred between Day 1 to Day 91 are reported under the Depot Buprenorphine treatment arm.
  Adverse events that occurred on the day of a hydromorphone challenge are also reported under the appropriate hydromorphone challenge treatment arm.
Groups:
- Depot Buprenorphine: Participants were treated with RBP-6000 300 mg in a single subcutaneous injection on Days 1 and 29.
Arm/Group | Depot Buprenorphine | Placebo Challenge | Hydromorphone 6 mg Challenge | Hydromorphone 18 mg Challenge
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 34/39 | 23/38 | 18/38 | 19/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Depot Buprenorphine (N=39) | Placebo Challenge (N=38) | Hydromorphone 6 mg Challenge (N=38) | Hydromorphone 18 mg Challenge (N=38)
Injection site erythema (General disorders) | 2 | 0 | 0 | 0
Injection site pruritis (General disorders) | 2 | 0 | 0 | 1
Local swelling (General disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 20 | 8 | 9 | 10
Sedation (Nervous system disorders) | 9 | 3 | 4 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 12 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 11 | 3 | 2 | 1
Vomiting (Gastrointestinal disorders) | 9 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 6 | 2 | 1 | 2
Anxiety (Psychiatric disorders) | 12 | 2 | 2 | 3
Abnormal dreams (Psychiatric disorders) | 4 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 1 | 2 | 0
Hot flush (Vascular disorders) | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.